CLINICAL TRIAL: NCT02939014
Title: A Phase 2, Single-Arm, Open-label Study of Brentuximab Vedotin in Chinese Patients With Relapsed/Refractory CD30-Positive Hodgkin Lymphoma (HL) or Systemic Anaplastic Large Cell Lymphoma (sALCL)
Brief Title: Brentuximab Vedotin in Chinese Participants With Relapsed/Refractory CD30-Positive Hodgkin Lymphoma (HL) or Systemic Anaplastic Large Cell Lymphoma (sALCL)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C25010; U1111-1184-1838 (Other: WHO)
Record Dates: First submitted 2016-10-18; First posted 2016-10-19 (Estimated); Results first posted 2019-09-06 (Actual); Last update posted 2021-02-24 (Actual); Status verified 2021-02

CONDITIONS: Hodgkin Disease; Lymphoma, Large-Cell, Anaplastic
Keywords: Drug therapy
MeSH Terms: conditions — Hodgkin Disease; Lymphoma, Large-Cell, Anaplastic | interventions — Brentuximab Vedotin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Brentuximab Vedotin 1.8 mg/kg (Experimental): Brentuximab vedotin 1.8 mg/kg, intravenous (IV) infusion on Day 1 of each 3-week cycle until the sooner of disease progression, unacceptable toxicity, or completion of 16 cycles.
  Interventions: Drug: Brentuximab Vedotin

INTERVENTIONS:
Drug: Brentuximab Vedotin — Brentuximab vedotin IV infusion

SUMMARY:
The purpose of this study is to evaluate the efficacy, safety and pharmacokinetics (PK) of brentuximab vedotin as a single agent in Chinese participants with relapsed/refractory CD30+ Hodgkin Lymphoma (HL) or Systemic Anaplastic Large Cell Lymphoma (sALCL).

DETAILED DESCRIPTION:
The drug being tested in this study is called brentuximab vedotin. This study will look at efficacy, safety and PK of brentuximab vedotin in Chinese participants with relapsed/refractory CD30+ HL or sALCL.

The study will enroll approximately 30 patients. Participants will receive:

• Brentuximab vedotin 1.8 mg/kg

All participants will be administered IV infusion on Day 1 each 3-week cycle until the sooner of disease progression, unacceptable toxicity, or completion of 16 cycles.

This multi-center trial will be conducted in China only. The overall time to participate in this study is 3.5 years. Participants will make multiple visits to the clinic, and will be followed for overall survival (OS) every 12 weeks until death, withdrawal of consent, 18 months after end of treatment (EOT) or study closure, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

1. Have histologically confirmed CD30+ hodgkin lymphoma (HL) or systemic anaplastic large cell lymphoma (sALCL). Immunohistochemistry or flow cytometry may be performed on either original diagnostic biopsy material or biopsy of relapsed disease, and pathology reports of CD30+ or their copies should be retained at the site.
2. With CD30+ HL or sALCL who have relapsed from or are refractory to previous treatments.
3. Fluorodeoxyglucose (FDG)- positron emission tomography (PET) positive and measurable disease of at least 1.5 cm in the longest diameter by computed tomography (CT), as assessed by the site.
4. Must have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
5. Suitable venous access for the study-required blood sampling, including pharmacokinetic (PK) sampling.
6. Must have the following required screening laboratory data. Participants must not have received recombinant granulocyte-colony stimulating factor (G-CSF) or platelet transfusion within 1 week before the screening hematology assessment.

   1. Absolute neutrophil count ≥1500/μL.
   2. Platelet count ≥75,000/μL.
   3. Serum bilirubin level ≤1.5 times the upper limit of the normal range (ULN).
   4. Serum creatinine level ≤1.5 times the ULN.
   5. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤2.5 times the ULN.
7. Survival for 3 or more months must be expected.

Exclusion Criteria:

1. With current diagnosis of primary cutaneous anaplastic large cell lymphoma (ALCL) (participants with other organ involvement who have transformed to sALCL are eligible).
2. With any active viral, bacterial, or fungal infection within 2 weeks before the first dose of brentuximab vedotin.
3. With cardiac failure categorized as Class III or IV according to the New York Heart Association criteria, uncontrolled coronary artery disease or uncontrolled arrhythmia despite of appropriate medical therapy, or a history of myocardial infarction within 6 months before the first dose of brentuximab vedotin.
4. With uncontrolled diabetes mellitus.
5. Peripheral neuropathy ≥Grade 2.
6. With a history of another malignancy that has not been in remission for at least 3 years. The following are exempt from the 3-year limit:

   1. Nonmelanoma skin cancer.
   2. Curatively treated localized prostate cancer.
   3. Cervical carcinoma in situ.
7. With known cerebral/meningeal disease (HL or any other etiology), including signs or symptoms of progressive multifocal leukoencephalopathy (PML).
8. With a positive result in the screening test for human immunodeficiency virus (HIV) antibody.
9. Known hepatitis B virus (HBV) surface antigen seropositive or positive hepatitis C virus (HCV) antibody. Note: participants who have positive HBV core antibody can be enrolled but must have an undetectable HBV viral load.
10. With a history of liver fibrosis or cirrhosis and clinical signs and symptoms indicating liver fibrosis or cirrhosis.
11. Have received autologous stem cell transplantation (auto-SCT) within 12 weeks before the first dose of brentuximab vedotin.
12. With history of allogeneic stem cell transplantation (allo-SCT).
13. Have received treatment for malignancies (including radiation, chemotherapy, and hormone therapy) within 4 weeks before the first dose of brentuximab vedotin and participants who have received treatment for malignancies with biologics (including molecular target drug) or radioisotopic therapy within 12 weeks before the first dose of brentuximab vedotin.
14. Have unresolved toxicity higher than Grade 1 (National Cancer Institute Common Terminology Criteria for Adverse Events [NCI CTCAE] version 4.03) attributed to any prior therapy/procedure (excluding alopecia or non-clinically significant and asymptomatic laboratory abnormalities).
15. Have received systemic corticosteroids at doses greater than the equivalent of 20 mg/day of prednisone within 1 week before the first dose of brentuximab vedotin.
16. Comorbid systemic illnesses or other severe concurrent disease which, in the judgment of the investigator, would make the participant inappropriate for entry into this study or interfere significantly with the proper assessment of the safety and toxicity of the prescribed regimens.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2016-11-07 (Actual); Primary Completion 2018-08-02 (Actual); Study Completion 2020-02-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director Clinical Science, Study Director — Takeda
Locations (7):
- China (7):
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - Sun Yat-san University Cancer Center, Guangzhou, Guangdong
  - Jiangsu Cancer Hospital, Nanjing, Jiangsu
  - Jiangsu Province People's Hospital, Nanjing, Jiangsu
  - The First Hospital of Jilin University, Changchun, Jilin
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda

REFERENCES:
- [Derived] Song Y, Guo Y, Huang H, Li W, Ke X, Feng J, Xu W, Miao H, Kinley J, Song G, Dai Y, Wang H, Zhu J. Phase II single-arm study of brentuximab vedotin in Chinese patients with relapsed/refractory classical Hodgkin lymphoma or systemic anaplastic large cell lymphoma. Expert Rev Hematol. 2021 Sep;14(9):867-875. doi: 10.1080/17474086.2021.1942831. Epub 2021 Aug 24. PMID 34275403

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 7 investigative sites in China. The study was conducted from 07 November 2016 to 3 February 2020.
Pre-assignment Details: Participants with a diagnosis of Relapsed/Refractory CD30-Positive Hodgkin Lymphoma (HL) or Systemic Anaplastic Large Cell Lymphoma (sALCL) were enrolled to receive brentuximab vedotin 1.8 mg/kg, intravenous (IV) infusion, Day 1 of every 3-week cycle.
Groups:
- Brentuximab Vedotin 1.8 mg/kg (HL): Brentuximab vedotin 1.8 mg/kg, IV, infusion on Day 1 of each 3-week cycle until the sooner of disease progression, unacceptable toxicity, or completion of 16 cycles in participants with Relapsed/Refractory CD30-Positive Hodgkin Lymphoma (HL).
- Brentuximab Vedotin 1.8 mg/kg (sALCL): Brentuximab vedotin 1.8 mg/kg, IV, infusion on Day 1 of each 3-week cycle until the sooner of disease progression, unacceptable toxicity, or completion of 16 cycles in participants with Relapsed/Refractory Systemic Anaplastic Large Cell Lymphoma (sALCL).
Period: Overall Study
Arm/Group | Brentuximab Vedotin 1.8 mg/kg (HL) | Brentuximab Vedotin 1.8 mg/kg (sALCL)
Started | 30 | 9
Completed (Completed included participants who completed 16 cycles of treatment with brentuximab vedotin and 18-months post-treatment follow-up.) | 25 | 6
Not Completed | 5 | 3
Not completed — Lost to Follow-up | 1 | 0
Not completed — Death | 4 | 3

BASELINE CHARACTERISTICS:
Population: Safety Population included all participants who had measurable lesions at baseline and received at least 1 dose of brentuximab vedotin.
Groups:
- Total: Total of all reporting groups
Arm/Group | Brentuximab Vedotin 1.8 mg/kg (HL) | Brentuximab Vedotin 1.8 mg/kg (sALCL) | Total
Number analyzed (Participants) | 30 | 9 | 39
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.9 (8.91) | 41.1 (15.28) | 34.0 (11.19)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 2 | 15
  Male | 17 | 7 | 24
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: Not Hispanic or Latino | 30 | 9 | 39
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Asian | 30 | 9 | 39
Region of Enrollment [Count of Participants; unit: Participants]
  China | 30 | 9 | 39

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR)
Description: ORR is defined as the percentage of participants who have achieved complete remission (CR)=disappearance of all evidence of disease or partial remission (PR)=regression of greater than or equal to 50% of measurable disease and no new site by end of treatment (EOT) per Cheson 2007 Revised Response Criteria for Malignant Lymphoma.
Time Frame: Baseline, at Cycles (each cycle was of 3 weeks) 2, 4, 7, 10, 13, and 16 during treatment until disease progression death or end of treatment (approximately 12 months)
Population: Modified Intent-to-Treat (mITT) Population included all participants who had measurable lesions at baseline and received at least 1 dose of brentuximab vedotin.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Brentuximab Vedotin 1.8 mg/kg (HL) | Brentuximab Vedotin 1.8 mg/kg (sALCL)
Number analyzed (Participants) | 30 | 9
percentage of participants | 70.0 [50.60 to 85.27] | 66.7 [29.93 to 92.51]

2. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: An Adverse Event (AE) is defined as any untoward medical occurrence in a clinical investigation participant administered a drug; it does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (eg, a clinically significant abnormal laboratory finding), symptom, or disease temporally associated with the use of a drug, whether or not it is considered related to the drug. A treatment-emergent adverse event (TEAE) is defined as an adverse event with an onset that occurs or worsens after receiving study drug.
Time Frame: First dose of study drug up to 30 days after last dose of study drug (approximately 12 months)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Brentuximab Vedotin 1.8 mg/kg (HL) | Brentuximab Vedotin 1.8 mg/kg (sALCL)
Number analyzed (Participants) | 30 | 9
Participants | 30 | 9

3. Primary Outcome: Number of Participants With Abnormal Clinical Laboratory Findings Reported as Adverse Events
Description: Clinical Laboratory tests included tests of Chemistry, Hematology and Urinalysis prespecified in the protocol. Abnormal laboratory values assessed by the investigator that lead to discontinuation or delay in treatment, dose modification, therapeutic intervention, or were considered by the investigator to be clinically significant changes from Baseline were recorded as Adverse Events. Neutropenia (pooled) includes preferred terms Neutropenia and Neutrophil count decreased.
Time Frame: First dose of study drug up to 30 days after last dose of study drug (approximately 12 months)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Brentuximab Vedotin 1.8 mg/kg (HL) | Brentuximab Vedotin 1.8 mg/kg (sALCL)
Number analyzed (Participants) | 30 | 9
Participants
  Alanine aminotransferase increased | 18 | 6
  Aspartate aminotransferase increased | 17 | 6
  Gamma-glutamyltransferase increased | 3 | 4
  Blood bilirubin increased | 0 | 2
  Reticulocyte count decreased | 9 | 2
  Reticulocyte count increased | 6 | 1
  Haemoglobin decreased | 1 | 1
  Reticulocyte percentage increased | 1 | 0
  White blood cell count decreased | 4 | 3
  Lymphocyte count decreased | 5 | 0
  Lymphocyte percentage decreased | 2 | 0
  Lymphocyte count increased | 0 | 1
  Lymphocyte percentage increased | 0 | 1
  Monocyte count increased | 0 | 1
  Neutrophil count increased | 0 | 1
  Neutrophil percentage decreased | 1 | 0
  White blood cell count increased | 0 | 1
  Platelet count decreased | 2 | 2
  Blood uric acid increased | 2 | 1
  Blood glucose increased | 1 | 1
  Blood albumin decreased | 0 | 1
  Protein total decreased | 0 | 1
  Blood creatinine increased | 1 | 1
  Blood urea decreased | 0 | 1
  Blood urea increased | 0 | 1
  Blood lactate dehydrogenase increased | 0 | 2
  Blood alkaline phosphatase increased | 0 | 1
  Blood cholesterol increased | 0 | 1
  Blood calcium decreased | 0 | 1
  Blood calcium increased | 0 | 1
  Blood chloride decreased | 0 | 1
  Blood phosphorus decreased | 0 | 1
  Blood potassium decreased | 0 | 1
  Blood triglycerides increased | 0 | 1
  Glucose urine present | 1 | 0
  Leukopenia | 15 | 2
  Anaemia | 12 | 3
  Hyperuricaemia | 4 | 2
  Hypertriglyceridaemia | 2 | 2
  Hypokalaemia | 3 | 2
  Blood creatine phosphokinase increased | 1 | 1
  Total bile acids increased | 0 | 2
  Alpha hydroxybutyrate dehydrogenase increased | 0 | 1
  Blood magnesium decreased | 0 | 1
  High density lipoprotein decreased | 0 | 1
  Hypercalcaemia | 0 | 1
  Hyperglycaemia | 1 | 0
  Hypoalbuminaemia | 0 | 1
  Hypocalcaemia | 0 | 1
  Hyponatraemia | 1 | 0
  Lipoprotein (a) increased | 0 | 1
  Low density lipoprotein increased | 0 | 1
  Monocytosis | 0 | 1
  Red blood cell sedimentation rate increased | 1 | 0
  Thrombocytopenia | 1 | 0
  Neutropenia (Pooled) | 19 | 5

4. Primary Outcome: Number of Participants With Abnormal Vital Signs Reported as Adverse Events
Description: Vital signs included blood pressure in the sitting position, pulse rate, axillary temperature and weight. Abnormal vital sign values considered by the investigator to be clinically significant were recorded as Adverse Events.
Time Frame: First dose of study drug up to 30 days after last dose of study drug (approximately 12 months)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Brentuximab Vedotin 1.8 mg/kg (HL) | Brentuximab Vedotin 1.8 mg/kg (sALCL)
Number analyzed (Participants) | 30 | 9
Participants
  Weight increased | 4 | 2
  Weight decreased | 1 | 2

5. Secondary Outcome: Complete Remission (CR) Rate
Description: CR rate is defined as the percentage of participants who have achieved CR by EOT. CR is defined as disappearance of all evidence of disease per Cheson 2007 Revised Response Criteria for Malignant Lymphoma.
Time Frame: Baseline, at Cycles (each cycle was of 3 weeks) 2, 4, 7, 10, 13, and 16 during treatment, and every 12 weeks during PFS follow-up period, until disease progression death or end of treatment (approximately 12 months)
Population: mITT Population included all participants who had measurable lesions at baseline and received at least 1 dose of brentuximab vedotin.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Brentuximab Vedotin 1.8 mg/kg (HL) | Brentuximab Vedotin 1.8 mg/kg (sALCL)
Number analyzed (Participants) | 30 | 9
percentage of participants | 20.0 [7.71 to 38.57] | 55.6 [21.20 to 86.30]

6. Secondary Outcome: Duration of Response (DOR)
Description: DOR is defined as the time between the first documentation of objective tumor response (CR or PR) and the first subsequent documentation of objective tumor progression or death due to any cause, whichever occurs first. CR is defined as disappearance of all evidence of disease. PR is defined as regression of greater than or equal to 50% of measurable disease and no new sites.
Time Frame: Up to 3.2 years
Population: mITT Population included all participants who had measurable lesions at baseline and received at least 1 dose of brentuximab vedotin. Only responders were analyzed for this outcome measure.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Brentuximab Vedotin 1.8 mg/kg (HL) | Brentuximab Vedotin 1.8 mg/kg (sALCL)
Number analyzed (Participants) | 21 | 6
months | 12.0 [4.37 to NA] — Data for upper limit of CI were not available as all participants were censored. | NA [1.41 to NA] — Data for upper limit of CI were not available as all participants were censored.

7. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS is defined as the time from the start of study treatment to the first documentation of objective tumor progression or to death due to any cause, whichever occurs first.
Time Frame: Up to 3.2 years
Population: as for outcome 5
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Brentuximab Vedotin 1.8 mg/kg (HL) | Brentuximab Vedotin 1.8 mg/kg (sALCL)
Number analyzed (Participants) | 30 | 9
months | 13.5 [6.77 to 17.81] | 23.2 [1.25 to NA] — Data for upper limit of CI was not available as all participants were censored.

8. Secondary Outcome: Overall Survival (OS)
Description: Overall survival is defined as the time from the start of treatment to the date of death.
Time Frame: Up to 3.2 years
Population: as for outcome 5
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Brentuximab Vedotin 1.8 mg/kg (HL) | Brentuximab Vedotin 1.8 mg/kg (sALCL)
Number analyzed (Participants) | 30 | 9
months | NA [NA to NA] — Data for Median and lower and Upper limit of CI was not available due to low number of participants with events. | NA [3.19 to NA] — Data for Median and lower and Upper limit of CI was not available due to low number of participants with events.

9. Secondary Outcome: B Symptom Resolution Rate
Description: B Symptom Resolution Rate is defined as the percentage of participants with lymphoma-related symptoms (B symptoms: fever, night sweats, or weight loss >10%) at baseline who achieved resolution of all B symptoms at any time during the treatment period.
Time Frame: Day 1 of each cycle (each cycle was of 3 weeks) up to 30 days after last dose of study drug (approximately 12 months)
Population: Participants from the mITT Population, all participants who had measurable lesions at baseline and received at least 1 dose of brentuximab vedotin, who had lymphoma-related B symptoms at baseline.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Brentuximab Vedotin 1.8 mg/kg (HL) | Brentuximab Vedotin 1.8 mg/kg (sALCL)
Number analyzed (Participants) | 2 | 2
percentage of participants | 50.0 [1.26 to 98.74] | 100.00 [15.81 to 100.00]

10. Secondary Outcome: Cmax: Maximum Observed Serum Concentration for Brentuximab Vedotin Antibody-drug Conjugate (ADC)
Time Frame: Cycles (each cycle was of 3 weeks) 1 and 2: Day 1 pre-dose and at multiple time points (up to 336 hours) post-dose
Population: Pharmacokinetic (PK)-evaluable Population includes participants with sufficient dosing and PK data to reliably estimate PK parameters as determined by the clinical pharmacologist.
Measure: Mean (Standard Deviation); unit: micrograms/milliliter (ug/mL)
Groups:
- Brentuximab Vedotin 1.8 mg/kg: Brentuximab vedotin 1.8 mg/kg, IV, infusion on Day 1 of each 3-week cycle until the sooner of disease progression, unacceptable toxicity, or completion of 16 cycles includes all participants.
Arm/Group | Brentuximab Vedotin 1.8 mg/kg
Number analyzed (Participants) | 39
micrograms/milliliter (ug/mL)
  Cycle 1 | 36.9504 (9.90360)
  Cycle 2 | 32.4341 (5.83197)

11. Secondary Outcome: Cmax: Maximum Observed Serum Concentration for Total Antibody (TAb)
Time Frame: Cycles (each cycle was of 3 weeks) 1 and 2: Day 1 pre-dose and at multiple time points (up to 336 hours) post-dose
Population: PK-evaluable Population includes participants with sufficient dosing and PK data to reliably estimate PK parameters as determined by the clinical pharmacologist.
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | Brentuximab Vedotin 1.8 mg/kg
Number analyzed (Participants) | 39
ug/mL
  Cycle 1 | 38.2293 (7.95483)
  Cycle 2 | 39.9859 (12.43445)

12. Secondary Outcome: Cmax: Maximum Observed Plasma Concentration for Monomethyl Auristatin E (MMAE)
Time Frame: Cycles (each cycle was of 3 weeks) 1 and 2: Day 1 pre-dose and at multiple time points (up to 336 hours) post-dose
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | Brentuximab Vedotin 1.8 mg/kg
Number analyzed (Participants) | 39
ug/mL
  Cycle 1 | 5.1623 (3.69893)
  Cycle 2 | 3.6218 (2.89331)

13. Secondary Outcome: Tmax: Time to Reach the Maximum Plasma Concentration (Cmax) for Brentuximab Vedotin ADC
Time Frame: Cycles (each cycle was of 3 weeks) 1 and 2: Day 1 pre-dose and at multiple time points (up to 336 hours) post-dose
Population: as for outcome 11
Measure: Median (Full Range); unit: days
Arm/Group | Brentuximab Vedotin 1.8 mg/kg
Number analyzed (Participants) | 39
days
  Cycle 1 | 0.0576 [0.031 to 0.221]
  Cycle 2 | 0.0528 [0.028 to 0.214]

14. Secondary Outcome: Tmax: Time to Reach the Maximum Serum Concentration (Cmax) for TAb
Time Frame: Cycles (each cycle was of 3 weeks) 1 and 2: Day 1 pre-dose and at multiple time points (up to 336 hours) post-dose
Population: as for outcome 11
Measure: Median (Full Range); unit: days
Arm/Group | Brentuximab Vedotin 1.8 mg/kg
Number analyzed (Participants) | 39
days
  Cycle 1 | 0.0653 [0.031 to 1.067]
  Cycle 2 | 0.0660 [0.028 to 0.972]

15. Secondary Outcome: Tmax: Time to Reach the Maximum Plasma Concentration (Cmax) for MMAE
Time Frame: Cycles (each cycle was of 3 weeks) 1 and 2: Day 1 pre-dose and at multiple time points (up to 336 hours) post-dose
Population: as for outcome 11
Measure: Median (Full Range); unit: days
Arm/Group | Brentuximab Vedotin 1.8 mg/kg
Number analyzed (Participants) | 39
days
  Cycle 1 | 2.0729 [1.031 to 6.991]
  Cycle 2 | 2.9785 [0.178 to 6.986]

16. Secondary Outcome: AUC(0-∞): Area Under the Serum Concentration-time Curve From Time 0 to Infinity for Brentuximab Vedotin ADC
Time Frame: Cycle (each cycle was of 3 weeks) 1: Day 1 pre-dose and at multiple time points (up to 336 hours) post-dose
Population: Participants from the PK-evaluable Populations, participants with sufficient dosing and PK data to reliably estimate PK parameters as determined by the clinical pharmacologist, with data available for analysis.
Measure: Mean (Standard Deviation); unit: day*ug/mL
Arm/Group | Brentuximab Vedotin 1.8 mg/kg
Number analyzed (Participants) | 38
day*ug/mL | 79.9951 (19.59116)

17. Secondary Outcome: AUC(0-∞): Area Under the Serum Concentration-time Curve From Time 0 to Infinity for TAb
Time Frame: Cycle (each cycle was of 3 weeks) 1: Day 1 pre-dose and at multiple time points (up to 336 hours) post-dose
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: day*ug/mL
Arm/Group | Brentuximab Vedotin 1.8 mg/kg
Number analyzed (Participants) | 39
day*ug/mL | 168.6618 (41.62840)

18. Secondary Outcome: AUC(0-∞): Area Under the Plasma Concentration-time Curve From Time 0 to Infinity for MMAE
Time Frame: Cycle (each cycle was of 3 weeks) 1: Day 1 pre-dose and at multiple time points (up to 336 hours) post-dose
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: day*ug/mL
Arm/Group | Brentuximab Vedotin 1.8 mg/kg
Number analyzed (Participants) | 39
day*ug/mL | 36.8625 (22.79816)

19. Secondary Outcome: Number of Participants With Antitherapeutic Antibodies (ATA) and Neutralizing Antitherapeutic Antibodies (nATA) to Brentuximab Vedotin
Description: Blood samples were collected to assess the immunogenicity of brentuximab vedotin (ATA development) using a laboratory test to determine ATA titers. Confirmed ATA-positive response was categorized as transient (defined as 1 or 2 post-baseline confirmed ATA-positive responses) and persistent (defined as more than 2 post-baseline confirmed ATA positive responses) and by nATA status. The number of participants in each baseline ATA and post-baseline ATA categories are reported.
Time Frame: Baseline, at Cycles (each cycle was of 3 weeks) 2, 4, 7, 10, 13, and 16 during treatment until disease progression, death or end of treatment (approximately 12 months)
Population: Immunogenicity Population included participants who received at least 1 dose of brentuximab vedotin and had ATA status assessment at baseline, and at least 1 postbaseline sample. Number analyzed is the number of participants with data available.
Measure: Count of Participants; unit: Participants
Arm/Group | Brentuximab Vedotin 1.8 mg/kg (HL) | Brentuximab Vedotin 1.8 mg/kg (sALCL)
Number analyzed (Participants) | 30 | 9
Participants
  Baseline ATA Negative | 29 | 9
  Baseline ATA Negative, ATA Negative: number analyzed (Participants) | 29 | 9
  Baseline ATA Negative, ATA Negative | 21 | 8
  Baseline ATA Negative, Transiently ATA Positive: number analyzed (Participants) | 29 | 9
  Baseline ATA Negative, Transiently ATA Positive | 7 | 1
  Baseline ATA Negative, Persistently ATA Positive: number analyzed (Participants) | 29 | 9
  Baseline ATA Negative, Persistently ATA Positive | 1 | 0
  Baseline ATA Negative, nATA Negative: number analyzed (Participants) | 8 | 1
  Baseline ATA Negative, nATA Negative | 0 | 0
  Baseline ATA Negative, nATA Positive: number analyzed (Participants) | 8 | 1
  Baseline ATA Negative, nATA Positive | 8 | 1
  Baseline ATA Positive | 1 | 0
  Baseline ATA Positive, ATA Negative: number analyzed (Participants) | 1 | 0
  Baseline ATA Positive, ATA Negative | 0 |
  Baseline ATA Positive, Transiently ATA Positive: number analyzed (Participants) | 1 | 0
  Baseline ATA Positive, Transiently ATA Positive | 0 |
  Baseline ATA Positive, Persistently ATA Positive: number analyzed (Participants) | 1 | 0
  Baseline ATA Positive, Persistently ATA Positive | 1 |
  Baseline ATA Positive, nATA Negative: number analyzed (Participants) | 1 | 0
  Baseline ATA Positive, nATA Negative | 0 |
  Baseline ATA Positive, nATA Positive: number analyzed (Participants) | 1 | 0
  Baseline ATA Positive, nATA Positive | 1 |

ADVERSE EVENTS:
Time Frame: All-Cause Mortality: up to 3.2 years; Serious and Other Adverse Events: First dose of study drug up to 30 days post last dose of study drug (up to 12 months)
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Brentuximab Vedotin 1.8 mg/kg (HL) | Brentuximab Vedotin 1.8 mg/kg (sALCL)
All-Cause Mortality (participants affected / at risk) | 4/30 | 3/9
Serious Adverse Events (participants affected / at risk) | 1/30 | 1/9
Other Adverse Events (participants affected / at risk) | 30/30 | 9/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Brentuximab Vedotin 1.8 mg/kg (HL) (N=30) | Brentuximab Vedotin 1.8 mg/kg (sALCL) (N=9)
Large intestine polyp (Gastrointestinal disorders) | 0 | 1
Lung infection (Infections and infestations) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Brentuximab Vedotin 1.8 mg/kg (HL) (N=30) | Brentuximab Vedotin 1.8 mg/kg (sALCL) (N=9)
Alanine aminotransferase increased (Investigations) | 18 | 6
Aspartate aminotransferase increased (Investigations) | 17 | 6
Gamma-glutamyltransferase increased (Investigations) | 3 | 4
Blood bilirubin increased (Investigations) | 0 | 2
Total bile acids increased (Investigations) | 0 | 2
Reticulocyte count decreased (Investigations) | 9 | 2
Reticulocyte count increased (Investigations) | 6 | 1
Haemoglobin decreased (Investigations) | 1 | 1
White blood cell count decreased (Investigations) | 4 | 3
Lymphocyte count decreased (Investigations) | 5 | 0
Lymphocyte percentage decreased (Investigations) | 2 | 0
Lymphocyte count increased (Investigations) | 0 | 1
Lymphocyte percentage increased (Investigations) | 0 | 1
Monocyte count increased (Investigations) | 0 | 1
Neutrophil count increased (Investigations) | 0 | 1
White blood cell count increased (Investigations) | 0 | 1
Weight increased (Investigations) | 4 | 2
Weight decreased (Investigations) | 1 | 2
Platelet count decreased (Investigations) | 2 | 2
Blood uric acid increased (Investigations) | 2 | 1
Retinol binding protein increased (Investigations) | 0 | 1
Blood glucose increased (Investigations) | 1 | 1
Blood albumin decreased (Investigations) | 0 | 1
Protein total decreased (Investigations) | 0 | 1
Blood creatinine increased (Investigations) | 1 | 1
Blood urea decreased (Investigations) | 0 | 1
Blood urea increased (Investigations) | 0 | 1
Blood creatine phosphokinase increased (Investigations) | 1 | 1
Alpha hydroxybutyrate dehydrogenase increased (Investigations) | 0 | 1
Blood lactate dehydrogenase increased (Investigations) | 0 | 2
Blood alkaline phosphatase increased (Investigations) | 0 | 1
Blood cholesterol increased (Investigations) | 0 | 1
High density lipoprotein decreased (Investigations) | 0 | 1
Lipoprotein (a) increased (Investigations) | 0 | 1
Low density lipoprotein increased (Investigations) | 0 | 1
Electrocardiogram abnormal (Investigations) | 0 | 1
Blood calcium decreased (Investigations) | 0 | 1
Blood calcium increased (Investigations) | 0 | 1
Blood chloride decreased (Investigations) | 0 | 1
Blood magnesium decreased (Investigations) | 0 | 1
Blood phosphorus decreased (Investigations) | 0 | 1
Blood potassium decreased (Investigations) | 0 | 1
Blood triglycerides increased (Investigations) | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 15 | 2
Anaemia (Blood and lymphatic system disorders) | 12 | 3
Neutropenia (Blood and lymphatic system disorders) | 19 | 5 — Neutropenia includes preferred terms Neutropenia and Neutrophil count decreased.
Monocytosis (Blood and lymphatic system disorders) | 0 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 9 | 2
Neuropathy peripheral (Nervous system disorders) | 0 | 2
Headache (Nervous system disorders) | 8 | 0
Hypoaesthesia (Nervous system disorders) | 4 | 2
Dizziness (Nervous system disorders) | 5 | 1
Diarrhoea (Gastrointestinal disorders) | 8 | 3
Nausea (Gastrointestinal disorders) | 8 | 0
Vomiting (Gastrointestinal disorders) | 4 | 1
Retching (Gastrointestinal disorders) | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 4 | 0
Flatulence (Gastrointestinal disorders) | 3 | 0
Dyspepsia (Gastrointestinal disorders) | 4 | 0
Abdominal pain upper (Gastrointestinal disorders) | 3 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 3 | 0
Abdominal discomfort (Gastrointestinal disorders) | 1 | 1
Gingival bleeding (Gastrointestinal disorders) | 0 | 1
Malaise (General disorders) | 6 | 1
Asthenia (General disorders) | 4 | 0
Pyrexia (General disorders) | 6 | 4
Pain (General disorders) | 3 | 0
Chest discomfort (General disorders) | 1 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 8 | 1
Rash (Skin and subcutaneous tissue disorders) | 3 | 2
Night sweats (Skin and subcutaneous tissue disorders) | 3 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 2 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 2 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 0
Papule (Skin and subcutaneous tissue disorders) | 0 | 1
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 9 | 2
Nasopharyngitis (Infections and infestations) | 1 | 1
Tonsillitis (Infections and infestations) | 0 | 1
Herpes zoster (Infections and infestations) | 2 | 1
Nail infection (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 4 | 2
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 2 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 3 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 0
Palpitations (Cardiac disorders) | 2 | 0
Insomnia (Psychiatric disorders) | 2 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In general, Investigators may publish clinical data after the earlier of (i) publication by the Sponsor or (ii) 12 months following the abandonment, early termination or database lock; provided a copy of the publication provided to Sponsor at least 30 days ahead of publication, the Sponsor's confidential information is removed as may be requested by Sponsor and Investigator defers publication for up to 60 days in the event Sponsor provides notice that it intends to file a patent application

DOCUMENTS (2):
  • Study Protocol (2016-04-20): https://cdn.clinicaltrials.gov/large-docs/14/NCT02939014/Prot_000.pdf
  • Statistical Analysis Plan (2018-08-30): https://cdn.clinicaltrials.gov/large-docs/14/NCT02939014/SAP_001.pdf